CLINICAL TRIAL: NCT00798330
Title: Pilot Study on Transient Bacteremia and Blood Stream Infections After Invasive Dental Procedures in Cancer Patients With Central Venous Catheters
Brief Title: Dental Study in Cancer Patients With Central Venous Catheters
Status: Completed | Type: Observational
Sponsor: Rajesh Lalla (Other)
Responsible Party: Sponsor-Investigator, Rajesh Lalla, Associate Professor, School of Dental Medicine, UConn Health
Organization: UConn Health (Other)
Other Study IDs: 09-059-2; 786-001
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cancer
Keywords: Cancer; Blood stream infections; Bacteremia; Dental procedure; Central venous catheters; Mediport; PICC line
MeSH Terms: conditions — Neoplasms; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients who are preparing to receive chemotherapy are asked to have their teeth cleaned before starting treatment as standard of care. This research study is being done to see if having dental cleaning increases the chances of bacteria from the mouth getting into the blood stream. It is also being done to see if these bacteria can cause blood stream infections in people who have a Central Venous Catheter (CVC),often called a "port" or a "PICC", placed for giving chemotherapy. It is a well-established fact that we introduce bacteria from the mouth into the bloodstream with activities of daily life including chewing, flossing and brushing teeth. This introduction of bacteria into the blood stream may cause bacteria to stick to the central venous catheter and serve as a source of infection when the immune system is weakened by cancer. The purpose of this research study is to see if we can find bacteria from mouth in blood that is drawn through the CVC, during, and after a dental cleaning procedure. This way, we will be able to assess whether or not this is a potential health risk to cancer patients.

ELIGIBILITY:
Inclusion criteria

* Patients willing and able to provide written informed consent for the study.
* Patients diagnosed with cancer and being treated at the University of Connecticut Health Center.
* Patients scheduled to receive or who have received a central venous catheter
* Patients who have at least one tooth.

Exclusion criteria

* Patients under the age of 18
* Patients who have received any antibacterial in the time period starting 48 hours before the dental cleaning. This includes systemic antibacterials and topical antibacterials in the oral cavity or at/through the CVC site. (Topical antibacterials at other sites are allowed; antifungal and antiviral agents in any form are allowed).
* Patients who plan to use antibacterials within the 24 hours after the procedure (until the final blood sample is obtained).
* Patients with a documented blood stream infection within 1 month prior to proposed dental cleaning.
* Patients with a clinically significant coagulation disorder or patients on warfarin.
* Patients who require antibiotic prophylaxis as per American College of Cardiology/American Heart Association (ACC/AHA) 2007 guidelines, namely;
* patients who have had a cardiac transplantation,
* incomplete cardiac valve repair,
* complete cardiac valve repair in last 6 months,
* prior history of infective endocarditis ,
* patients with a prosthetic cardiac valve.
* Patients with any other condition which might preclude participation in the opinion of the patient's physician(s) or the study PI's.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer outpatients with central venous catheters (Medport or PICC lines)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of transient bacteremia and established blood-stream infections (BSIs) by oral microorganisms in cancer patients with CVCs after an invasive dental procedure | Two days, 1 month, 6 months
  Blood cultures drawn before dental cleaning, 20 minutes after starting procedure, 30 minutes after finishing the procedure and at 24 hours after starting the procedure. Records reviewed at one month and six months post procedure for bloodstream or central venous catheter infection.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh V Lalla, DDS, Ph.D, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Usmani S, Choquette L, Bona R, Feinn R, Shahid Z, Lalla RV. Transient bacteremia induced by dental cleaning is not associated with infection of central venous catheters in patients with cancer. Oral Surg Oral Med Oral Pathol Oral Radiol. 2018 Apr;125(4):286-294. doi: 10.1016/j.oooo.2017.12.022. Epub 2018 Jan 11. PMID 29428697
- See also: Publication describing results of this study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5944361/